CLINICAL TRIAL: NCT02204046
Title: A Phase I Biodistribution Study With 186 Re-labelled Humanised Monoclonal Antibody BIWA 4, in Patients With Adenocarcinoma of the Breast
Brief Title: Biodistribution Study With 186 Re-labelled Humanised Monoclonal Antibody BIWA 4 in Patients With Adenocarcinoma of the Breast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1170.2
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — monoclonal antibody BIWA 4

ARMS (1):
- BIWA 4 (Experimental): Generic Name: Bivatuzumab
  186Re-labelled humanised monoclonal antibody BIWA 4
  Interventions: Drug: BIWA 4

INTERVENTIONS:
Drug: BIWA 4

SUMMARY:
The primary objectives of this study were to assess the safety and tolerability of intravenously (i.v.) administered 186Rhenium (186Re)-labelled bivatuzumab and to investigate the biodistribution and pharmacokinetics of 186Re-labelled bivatuzumab in patients with adenocarcinoma of the breast

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or cytological confirmation of a primary adenocarcinoma of the breast
* Patients destined for tumour extirpation or mastectomy
* Patients over 18 years of age
* Patients younger than 80 years of age
* Patients who had given 'written informed consent'
* Patients with a life expectancy of at least 3 months
* Patients with a good performance status: Karnofsky > 60

Exclusion Criteria:

* Life-threatening infection, allergic diathesis, organ failure (bilirubin > 30µmol/l and/or creatinine > 150 µmol/l) or evidence of a recent myocardial infarction on ECG or unstable angina pectoris
* Pre-menopausal women (last menstruation <= 1 year prior to study start)

  * Not surgically sterile (hysterectomy, tubal ligation) and
  * Not practicing acceptable means of birth control, (or not planned to be continued throughout the study). Acceptable methods of birth control include oral, implantable or injectable contraceptives
* Women with a positive serum pregnancy test at baseline
* White blood cell count < 3000/mm³, granulocyte count < 1500/mm³ or platelet count < 100000/mm³. Details of prior chemotherapy or radiotherapy had to be known
* Hematological disorders, congestive heart failure, bronchial asthma, alimentary or contact allergy, severe atopy or allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2000-01; Primary Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 6 weeks after infusion
Number of patients with abnormal changes in laboratory parameters | up to 6 weeks after infusion
Number of patients with clinically significant changes in vital signs | up to 6 weeks after infusion
Presence of Human-Anti-Human-Antibody (HAHA) | up to 6 weeks after infusion
Uptake of 186Re-labelled hMAb BIWA 4 in tumour and normal tissue samples | up to 72 hours after infusion
  Assessment of biodistribution by radioscintigraphy expressed as low, medium or high
AUC0-∞ (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 240 hours after infusion
Cmax (Maximum measured concentration of the analyte in plasma) | up to 240 hours after infusion
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 240 hours after infusion
t½ (Terminal half-life of the analyte in plasma) | up to 240 hours after infusion
MRT (Mean residence time of the analyte in the body) | up to 240 hours after infusion
Vss (Apparent volume of distribution under steady state conditions) | up to 240 hours after infusion
Vz (Apparent volume of distribution during the terminal phase) | up to 240 hours after infusion
CL (Total body clearance) | up to 240 hours after infusion
Actual uptake of 186Re-labelled hMAb BIWA 4 in tumour and normal tissue samples | at 72 hours after infusion
  expressed as %ID/kg
Uptake of 186Re-labelled hMAb BIWA 4 in tumour and normal tissue samples | after surgery on day 8
  Biodistribution assessed from biopsy sample as percentage of the injected dose per kg tissue (%ID/kg)